CLINICAL TRIAL: NCT05897814
Title: Evaluation of M-mode Ultrasonography for Epidural Catheter Identification, and Correct Placement, in Obstetric Anesthesia
Brief Title: M-mode Ultrasonography for Epidural Catheter Identification and Confirmation of Correct Catheter Position
Acronym: ETEMERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230314; 2023-A00076-39 (Other: IDRCB Number)
Record Dates: First submitted 2023-05-11; First posted 2023-06-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Epidural Analgesia for Labour and Delivery
Keywords: Epidural anesthesia; Localization of the epidural analgesia catheter; Lumbar neuraxial ultrasound; Color Doppler mode; M-mode ultrasonography; Obstetric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parturients (Experimental): Adult patients admitted to the delivery room of Necker-Enfants Malades hospital maternity with an epidural catheter.
  Interventions: Other: Location of the epidural analgesia catheter

INTERVENTIONS:
Other: Location of the epidural analgesia catheter — Research of the location of the epidural analgesia catheter using M-mode and color Doppler (cD) ultrasonography.

SUMMARY:
In France, 80% of women choose epidural analgesia for delivery and birth. The localization of the epidural space is classically achieved by loss of resistance to saline. This blind technique means the passage of the needle through the ligamentum flavum. However, epidural analgesia failure has been reported in 27-32% of cases.

Currently, lumbar neuraxial ultrasound has become a valuable tool facilitating the placement of an epidural catheter. Although lumbar neuraxial ultrasound has been the source of many studies, few have focused on its use to confirm the exact location of the epidural catheter in the epidural space.

In the Pediatric and Obstetric Anesthesia-Resuscitation Department of the Necker-Enfants Malades Hospital, pre procedural lumbar neuraxial ultrasound for epidural anesthesia is a regular practice.

The objective of this study is to evaluate the ability of M-mode (M-m) and color Doppler (cD) ultrasonography to identify the epidural catheter position for parturients in the delivery room.

DETAILED DESCRIPTION:
In France, 80% of women choose epidural analgesia for delivery and birth. The localization of the epidural space is classically achieved by loss of resistance to saline. This blind technique means the passage of the needle through the ligamentum flavum. However, epidural analgesia failure has been reported in 27-32% of cases.

Currently, lumbar neuraxial ultrasound has become a valuable tool facilitating the placement of an epidural catheter. Although lumbar neuraxial ultrasound has been the source of many studies, few have focused on its use to confirm the exact location of the epidural catheter in the epidural space.

Indeed, only 2 retrospective studies have described this strategy on cohorts with small numbers of adult patients. One demonstrated in a mixed population the possible localization of the epidural analgesia catheter using color Doppler (cD) mode (67.5% of cases) and M-mode (M-m) ultrasonography (M-m) (75%). Only one study identified the position of the epidural catheter in the obstetric context due to the cD mode ; with a low rate of visualization (37.1% of cases).

In the Pediatric and Obstetric Anesthesia-Resuscitation Department of the Necker-Enfants Malades Hospital, pre procedural lumbar neuraxial ultrasound for epidural anesthesia is a regular practice.

The objective of this study is to evaluate the ability of the M-m and cD mode to identify proper catheter placement in parturients in the delivery room.

ELIGIBILITY:
Inclusion Criteria:

* Adult women admitted to the delivery room for a vaginal delivery with an epidural analgesia.
* Written informed consent.
* French speaking patient.

Exclusion Criteria:

* Patient with a contraindication to neuraxial analgesia.
* Visual Analogue Scale score >7 at epidural analgesia pose.
* No health insurance.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
Success rate of epidural catheter localisation in M-mode (M-m) ultrasonography | Day 0
  The location of the epidural catheter is based on the visualization of the "beach and sea" sign with injection of the analgesic solution through the epidural catheter into the epidural space.

SECONDARY OUTCOMES:
Success rate of epidural catheter localisation in color Doppler (cD) ultrasonography | Day 0
  The localization of the epidural catheter is based on the visualization of a blue and red mosaic with the injection of the analgesic solution through the epidural catheter in the epidural space.
Risk factors associated with location failure in M-m et cD mode | 14 months
  Description of the risk factors associated with catheter localization failure using M-mode (M-m) and color Doppler (cD) mode.
Best neuraxial ultrasound view to locate the epidural analgesia catheter with M-mode (M-m) and color Doppler (cD) mode | 14 months
  Determine the best neuraxial ultrasound view to locate the epidural catheter with M-mode (M-m) and color Doppler (cD) mode.
Evaluate the effectiveness of epidural analgesia when the catheter is considered in the epidural space by lumbar neuraxial ultrasound | Day 0
  Evaluate the percentage of epidurals having had a symmetrical sensory level > D10 when the epidural catheter is considered in the epidural space by lumbar neuraxial ultrasound.
  The epidural analgesia rate with a sensory level >D10 is determined 30 min after epidural analgesia application thanks to a sensitive test.
Duration of neuraxial ultrasound's research to determine the localization of epidural analgesia catheter | Day 0
  Evaluate the time required in minutes to confirm the correct positioning of the epidural analgesia catheter using M-m and cD mode.
Assess operator satisfaction with M-mode (M-m) and color Doppler (cD) to locate the epidural catheter | Day 0
  Operator satisfaction score with M-mode (M-m) and color Doppler (cD) to locate the epidural analgesia catheter with a numerical scale from 0 to 10.
Evaluate the satisfaction of parturients in terms of comfort during the lumbar neuraxial ultrasound to identify the epidural catheter | Day 0
  Evaluate the satisfaction of parturients in terms of comfort during the lumbar neuraxial ultrasound to identify the epidural catheter with a numerical scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Lauranne Ossé, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Hawa Keita-Meyer, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanhaesebrouck A, Vilain A, Rey S, Fresson J. Les maternités en 2016: résultats de l'enquête nationale périnatale (ENP). Revue d'Épidémiologie et de Santé Publique. 2018;66:S54
- [Background] Sicard JA, Forestier J. Radiographic method for exploration of the extradural space using lipidol. Rev Neurol. 1921;28:1264
- [Background] Perlas A, Chaparro LE, Chin KJ. Lumbar Neuraxial Ultrasound for Spinal and Epidural Anesthesia: A Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):251-60. doi: 10.1097/AAP.0000000000000184. PMID 25493689
- [Background] Elsharkawy H, Sonny A, Govindarajan SR, Chan V. Use of colour Doppler and M-mode ultrasonography to confirm the location of an epidural catheter - a retrospective case series. Can J Anaesth. 2017 May;64(5):489-496. doi: 10.1007/s12630-017-0819-y. Epub 2017 Jan 10. PMID 28074426
- [Background] Riveros-Perez E, Albo C, Jimenez E, Cheriyan T, Rocuts A. Color your epidural: color flow Doppler to confirm labor epidural needle position. Minerva Anestesiol. 2019 Apr;85(4):376-383. doi: 10.23736/S0375-9393.18.13175-0. Epub 2018 Nov 22. PMID 30482003